CLINICAL TRIAL: NCT01203670
Title: Renal and Digestive Tolerance of a Food Supplement, Phytalgic, in Elderly Volunteers - A Multicentric Open Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phythea (Industry)
Responsible Party: Pr. Nicholas MOORE, Département de pharmacologie Clinique - Université Victor Segalen Bordeaux 2 - Centre hospitalier universitaire de Bordeaux
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PHYTHEA-e437-950
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Renal Tolerance; Digestive Tolerance
Keywords: Glomerular filtration rate (GFR); Aspartate Amino Transferase (ASAT); Alanine Amino transferase (ALAT); gamma Glutamyl transpeptidase (gamma GT); Lipase; Amylase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Soft capsules of Phytalgic (Experimental): Phytalgic is a food supplement. Its galenic form is soft capsule.
  Interventions: Dietary Supplement: Phytalgic

INTERVENTIONS:
Dietary Supplement: Phytalgic — Volunteers have to take three soft capsules per day, one in the morning and two in the evening.

SUMMARY:
The aim of the study is to evaluate renal and digestive tolerance of a food supplement, phytalgic, on elderly volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old minimum
* Satisfying general health judged by principal investigator
* Pain and /or stifness associated with arthritis
* Regular used of analgesics and/or non-steroidal anti-inflammatory drugs (NSAIDs)
* Digestive tolerance biomarkers

  1. ASAT : Men < 150 UI/L - Women < 100 UI/L
  2. ALAT : Men < 180 UI/l - Women < 130 UI:l
  3. Gamma GT Men < 180 UI/l - Gamma GT Women < 100 UI/l
  4. Amylase < 250 UI/l
  5. Lipase < 750 UI/l
* Renal tolerance biomarker: Glomerular filtration rate (GFR)superior or equal to 60 mL /min / 1.73m3 - calculated with the "Modification of the Diet in Renal Diseases" formula

Exclusion Criteria:

* Inflammatory arthritis
* Allergy to any constituents of the study drug
* Types 2 diabetes
* Not legally fit to participate
* Any treatment able to modify determined biological parameters

Ages: 70 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Renal tolerance by Glomerular filtration rate (GFR) determination; Digestive tolerance by Aspartate Amino transferase (ASAT), Alanine Amino Transferase (ALAT), gamma Glutamyl Transpeptidase (gamma GT), lipase and amylase determination | 168 days

SECONDARY OUTCOMES:
Quality of life determined by Western Ontario and McMaster universities (WOMAC)Visual Analogue Scale(VAS) | 168 days

CONTACTS AND LOCATIONS:
Overall Officials: Alain JACQUET, MD, Principal Investigator — Département de pharmacologie Clinique - Université Victor Segalen Bordeaux 2 - Centre Hospitalo-Universitaire de Bordeaux
Locations (1):
- Département de Pharmacologie Clinique - Université Victor Segalen Bordeaux 2 - CHU de Bordeaux, Bordeaux, France